CLINICAL TRIAL: NCT06318715
Title: A Comparison of a Modified Deep Extubation to Standard Awake Extubation for Decreasing Operating Room Time: a Randomized Controlled Trial
Brief Title: Modified Deep Extubation vs. Standard Awake Extubation
Acronym: mDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0009-A
Record Dates: First submitted 2024-02-02; First posted 2024-03-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Extubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- modified deep extubation (Experimental): This modified deep extubation (mDE) occurs while the patient is still anaesthetized but at a lower dose of anaesthetic gas than previously described, and balanced with long acting opioids to attenuate the airway reaction.
  Interventions: Procedure: modified deep extubation (mDE)
- standard awake extubation (Experimental): awake extubation (AE) is still considered the standard practice.
  Interventions: Procedure: standard awake extubation

INTERVENTIONS:
Procedure: modified deep extubation (mDE) — The proposed study is to compare a modified DE technique, which is regularly used for low-risk patients by staff anesthesiologists at our institution, to a standard awake extubation.
  Arms: modified deep extubation
Procedure: standard awake extubation — awake extubation (AE) is still considered the standard practice.
  Arms: standard awake extubation

SUMMARY:
The proposed study is to compare a modified DE technique, which is regularly used for low-risk patients by staff anesthesiologists at our institution, to a standard awake extubation. This modified deep extubation (mDE) occurs while the patient is still anaesthetized but at a lower dose of anaesthetic gas than previously described, and balanced with long acting opioids to attenuate the airway reaction. As previously stated, the literature shows that the risks of DE are equivalent to those of regular AE practice. Our hypothesis is that mDE will shorten the time from the end of the surgery (completion of last stitch) to the moment the patient is ready to leave the OR by at least 5 minutes when compared to standard AE practice.

DETAILED DESCRIPTION:
Study type Randomized Controlled Trial comparing two extubation strategies for low-risk airway elective patients undergoing general anesthesia.

Population

* Inclusion criteria ASA I-III patients, scheduled for laparoscopic surgery under general anesthesia.
* Exclusion criteria

  * High-risk patients

    * Documented difficult airway during intubation or developed intraoperatively.
    * Full stomach
    * Pregnant women
    * Emergency surgery
    * BMI>30
    * Intraoperative bleeding leading to transfusion
  * Use of remifentanil during extubation
  * Requirement for prone position for surgical approach (i.e., spine surgery, anal fistulectomy, tumor resection of the back, etc)
  * Absolute indication for awake or deep extubation
  * Use of opioids in chronic pain patients

Procedures Patients that are potential candidates for the study will be selected according to inclusion and exclusion criteria when they undergo assessment on the Pre-Admission Unit (PAU). They will be selected from the PAU assessment list the day before the appointment by the research assistant. For both in person and phone interviews, the PAU personnel (nurse or anesthesiologist) will briefly introduce the patient to the study, and if the patient is interested in participating, the research assistant will approach them with detailed information and a hard-copy leaflet (or an email copy for a phone interview, if the patient agrees) regarding the study.

Informed consent to participate in the study will be taken by the research assistant on the day of surgery during the anesthesia assessment in the preoperative area. Patients will be randomized to either the AE or mDE group. Randomization will be performed in advance, using a computer-generated program and the participant assigned number. The patient and the research assistant will be blinded to the study group allocation. A study investigator, who will know the allocation of the patient, will assign the patient to the anesthesiologists that will provide the anesthesia and perform the extubation process according to group allocation. The anesthesiologists that are part of the research team will perform the extubation in the mDE group, and other attending anesthesiologists will perform their standard awake extubation in the AE group.

In the AE group, the attending anesthesiologist will perform the extubation according to the standard practice as follows:

1. Sevoflurane (anesthetic gas) will be reduced and the ventilator will be set up to wean patients from mechanical support using the anesthesiologist's method of preference.
2. Long-acting opioid (morphine or hydromorphone) will be given as per their clinical judgement.
3. Reversal of neuromuscular block will be performed in all patients and confirmed by a nerve stimulator Train of Four (TOF) ratio of > 0.9, which is the standard practice in patients receiving muscle relaxants as per the last clinical guidelines.
4. Oral suctioning will be performed.
5. Patients will be extubated once they are able to obey a verbal command of "open your eyes".
6. If needed, relief of airway obstruction will be performed at the discretion of the attending anesthesiologist using means such as an oral airway, or a jaw-thrust maneuver.

In the mED group, the attending anaesthesiologist who is familiar with the mDE technique will use the following protocol:

1. Towards the end of the surgery, sevoflurane will be set at an end-tidal concentration (ET%) of 0.7 MAC, the ventilator will be set to pressure support mode, and the patient will be allowed to breathe spontaneously.
2. A low dose of long-acting opioid (morphine 0.05 mg/kg or hydromorphone 0.01 mg/kg) will be given before the end of the surgery, according to the anesthesiologist's criteria.
3. Reversal of neuromuscular block will be performed in all patients and confirmed by a nerve stimulator TOF ratio of > 0.9, which is the standard practice in patients receiving muscle relaxants as per the last clinical guidelines).17
4. Oral suctioning will be performed while the patient is on Sevoflurane 0.7 MAC. The use of oral airway to avoid airway obstruction will be at the anesthesiologist discretion.
5. Ventilation support will be changed to the spontaneous mode after confirming an adequate respiratory drive on pressure support mode. Sevoflurane will then be stopped at the time of the last surgical stitch, and the fresh gas flow (FGF) with FiO2 1.0 will be adjusted at 18 litres/minute to optimize gas washout.
6. The patient will be extubated on spontaneous ventilation as soon as the ET% of sevoflurane drops to 0.4 MAC, once they achieve a minimum tidal volume of more than 3 millilitres per kilogram of ideal body weight and a respiratory rate of 8-12 breaths per minute, while they are still anesthetized under the effect of sevoflurane.
7. If needed, relief of airway obstruction will be performed at the discretion of the attending anesthesiologist by using means such as an oral airway, or a jaw-thrust maneuver.

During the patient care, the research assistant will record the events and times correlating to the primary and secondary outcomes by direct observation of the extubation process. The patient will also be interviewed by the research assistant in PACU regarding their experience with the recovery process once they are fully awake and ready to be transferred to the ward or discharged home. The patient will be blind to the allocation of the study group until the end of interview. If any problems occur during the extubation process, the patient will be debriefed by the attending anesthesiologist as regularly done in these cases regardless of study participation.

In case the patient was considered as a difficult intubation at the beginning of the case, or that the patient develops respiratory or hemodynamic instability, they would be excluded from the study and the extubation process will be carried out according to the attending anesthesiologist's clinical judgment.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* laparoscopic surgery under general anesthesia

Exclusion Criteria:

* High-risk patients:

  * Documented difficult airway during intubation or developed intraoperatively.
  * Full stomach
  * Pregnant women
  * Emergency surgery
  * BMI>30
  * Intraoperative bleeding leading to transfusion
* Use of remifentanil during extubation
* Requirement for prone position for surgical approach (i.e., spine surgery, anal fistulectomy, tumor resection of the back, etc)
* Absolute indication for awake or deep extubation
* Use of opioids in chronic pain patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time from the end of the surgery to leaving the OR | Time from the end of the surgery (completion of the last stitch) to the time the patient is ready to safely leave the OR
  Time from the end of the surgery (completion of the last stitch) to the time the patient is ready to safely leave the OR (defined as the moment when the patient breaths spontaneously with SpO2 > 97 % while receiving oxygen by a facial mask at 6-8 L/min, with normal chest wall movement, no airway obstruction and the presence of ETCO2 waveform).

SECONDARY OUTCOMES:
Time from the end of the surgery to extubation | Time from the end of the surgery (completion of the last stitch) to the moment of extubation
  Time from the end of the surgery (completion of the last stitch) to the moment of extubation (representing the period of extubation that is part of the surgical time).
Time from the end of the surgery to discharge from PACU | Time from the end of the surgery to the moment the patient is ready to be discharged from PACU
  Time from the end of the surgery to the moment the patient is ready to be discharged from PACU (Aldrete score greater or equal than 9) as per institutional protocol
oral airway | from intubation to extubation during the surgery/procedure
  Incidence of usage of oral airway.
jaw-thrust maneuver | from intubation to extubation during the surgery/procedure
  Incidence of performance of jaw-thrust maneuver and time of usage.
hypertension | During the first 5 minutes after extubation
  Incidence of hypertension defined as blood pressure higher than 20% of the baseline during the first 5 minutes after extubation.
breath holding | day 0
  Incidence of breath holding for more than 30 seconds after extubation.
bag-mask ventilation | day 0
  Incidence of need for bag-mask ventilation after extubation.
coughing | During the first minute after extubation.
  Incidence of coughing during the first minute after extubation.
bucking | During the first minute after extubation.
  Incidence of bucking during the first minute after extubation.
laryngospasm | day 0
  Incidence of laryngospasm (as identified by the attending anesthesiologist).
treat laryngospasm | day 0
  Usage of measures to treat laryngospasm (positive pressure ventilation, 0.5 mg/kg of iv propofol, or 0.3 mg/Kg of succinylcholine, or reintubation).
desaturation | day 0
  Incidence of desaturation (SPO2 less than 92%) after extubation.
reintubation | day 0
  Incidence of reintubation.2
Patient's experience | day 0
  Patient's experience using a questionnaire
BP | Just before extubation, and 1 minute and 5 minutes after extubation.
  Systolic and Diastolic Blood Pressure
HR | Just before extubation, and 1 minute and 5 minutes after extubation.
  Hear rate
EtCO2 | Just before extubation, and 1 minute and 5 minutes after extubation.
  End-tidal carbon dioxide
SaO2 | Just before extubation, and 1 minute and 5 minutes after extubation.
  oxygen saturation level
Sevorane MAC | Just before extubation, and 1 minute and 5 minutes after extubation.
  minimum alveolar concentration (MAC) for sevoflurane

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia Mount Sinai Hospital, Toronto, Ontario, Canada